CLINICAL TRIAL: NCT03418844
Title: Living After a Rare Cancer of the Ovary: Chronic Fatigue, Quality of Life and Late Effects of Chemotherapy
Acronym: VIVROVAIRE TR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Collaborators: ARCAGY/ GINECO GROUP (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: VIVROVAIRE TR
Record Dates: First submitted 2018-01-15; First posted 2018-02-01 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-08

CONDITIONS: Germ Cell Tumor; Sex Cord Stromal Tumor; Malignant Non-epithelial Ovarian Tumors
MeSH Terms: conditions — Neoplasms, Germ Cell and Embryonal; Sex Cord-Gonadal Stromal Tumors | interventions — Quality of Life

STUDY DESIGN:
Intervention Model Description: Patients and healthy volunteers will complete several self-questionnaires on living conditions and quality of life. Patients will also perform a cardiac, pulmonary, auditory and biological assessment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Interest group (patients treated with chemotherapy) (Other): Patients will complete several self-questionnaires on living conditions and quality of life. They will also perform a cardiac, pulmonary, auditory and biological assessment
  Interventions: Other: Self-questionnaires of living conditions and quality of life; Diagnostic Test: Cardiac, pulmonary, auditory and biological assessment
- Patient control group (patients not treated with chemotherapy) (Other): Patients will complete several self-questionnaires on living conditions and quality of life. They will also perform a cardiac, pulmonary, auditory and biological assessment
  Interventions: Other: Self-questionnaires of living conditions and quality of life; Diagnostic Test: Cardiac, pulmonary, auditory and biological assessment
- Healthy volunteers (Other): Healthy volunteers will complete several self-questionnaires on living conditions and quality of life.
  Interventions: Other: Self-questionnaires of living conditions and quality of life

INTERVENTIONS:
Other: Self-questionnaires of living conditions and quality of life — Patients will complete self-questionnaires of living conditions and quality of life (MFI-20, FACT-G/FACT-O, FACT/COG-NTX, FACT-Cog, HADS, Insomnia Severity Index , International Physical Activity Questionnaire)
Diagnostic Test: Cardiac, pulmonary, auditory and biological assessment — Patients will perform :
  * Cardiac assesments (ECG, Carotid and humeral Doppler ultrasound, Trans-thoracic echocardiography 2D and 3D)
  * Pulmonary and auditory assesment ( Respiratory Functional Exploration, Tonal audiogram)
  * Blood tests
  Arms: Interest group (patients treated with chemotherapy); Patient control group (patients not treated with chemotherapy)

SUMMARY:
While they are documented in patients in remission of testicular cancer, the sequelae of chemotherapy and the impact of the disease and its treatments on the living conditions and QoL of women in remission of rare ovarian cancer remain poorly explored.

The coordinator therefore propose a national 2-step case-control study to evaluate 1) chronic fatigue and QoL and 2) chemotherapy-related sequelae in adult patients in remission of surgery-treated TGMO or TSCS (conservative or not) supplemented with chemotherapy

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years;
* Patient with an ovarian malignant germ cell tumor (TGMO) or a stroma tumor and / or sex cords (TSCS) treated optimally;
* Patient who has had surgery and chemotherapy (interest group) or only a surgery (control group);
* Patient in remission more than 2 years after the end of the initial treatment;
* Relapse authorized if remission more than 2 years after the end of the treatment;
* Patient with no other cancers (with the exception of basal cell skin carcinomas, in situ cancers of the breast and cervix);
* Patient having signed his consent to participate

Exclusion Criteria:

* Pregnant or breastfeeding woman;
* Psychiatric pathology that may disrupt the course of the study or prevent the interpretation of results;
* Person deprived of liberty;
* Major subject to a legal protection measure or unable to express his consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 268 (Estimated)
Dates: Start 2018-05-07 (Actual); Primary Completion 2021-07-13 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The chronic fatigue by questionnaires | 2 years after surgery
The late sequelae of chemotherapy, particularly cardiovascular and pulmonary disorders, in adult patients in remission of a rare cancer of the ovary treated by surgery, supplemented or not by chemotherapy. | 2 years after surgery
The quality of life by questionnaires | 2 years after surgery

SECONDARY OUTCOMES:
The fertility monitoring by questionnaires | 2 years after surgery
The symptoms of menopause by questionnaires | 2 years after surgery
Theimpact of cancer and its treatments on the trajectory and professional situation by questionnaires(access to work, professional ambition, financial situation ...); | 2 years after surgery
The parental projects by age (≤ 45 years) by questionnaires | 2 years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Florence JOLY, Principal Investigator — Centre François Baclesse
Locations (19):
- France (19):
  - HEGP, Paris, Paris
  - Centre Paul Papin, Angers
  - CHU Besançon Jean MINJOZ, Besançon
  - Institut Bergonié, Bordeaux
  - CH Fleyriat, Bourg-en-Bresse
  - Centre François Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Léon Berard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Centre Catherine de Sienne, Nantes
  - Institut de Cancérologie de l'Ouest, Nantes
  - GH Cochin Broca Hôtel-Dieu, Paris
  - Hôpital Diaconesses-Croix St Simon, Paris
  - Institut Curie,, Paris
  - Institut Gustave Roussy, Paris
  - CHU Poitiers, Poitiers
  - Institut Jean Godinot, Reims
  - Institut Rennais de Cancérologie, Rennes
  - CHRU Stasbourg Hôpital Civil, Strasbourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dubot C, Ray-Coquard I, Lequesne J, Pautier P, Renaud T, Selle F, Berton-Rigaud D, Frank S, De La Motte Rouge T, Kalbacher E, Provansal M, Blonz C, Orfeuvre H, Alexandre J, Augereau P, Nadeau C, Kurtz JE, Hanvic B, Fresneau B, Ahmed-Lecheheb D, Christy F, Grellard JM, Clarisse B, Gernier F, Joly F. Long-term quality of life in non-epithelial ovarian cancer survivors: TMRG-GINECO-Vivrovaire rare tumors case-control study. BMC Med. 2025 Dec 12;24(1):34. doi: 10.1186/s12916-025-04540-x. PMID 41382138